CLINICAL TRIAL: NCT02757040
Title: Combination of Ibrutinib and As2O3 in the Treatment of CLL
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University People's Hospital (Other)
Collaborators: Beijing Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ibrutinib combined study
Record Dates: First submitted 2016-04-17; First posted 2016-04-29 (Estimated); Last update posted 2016-04-29 (Estimated); Status verified 2016-04

CONDITIONS: Leukemia, Lymphocytic, Chronic, B-Cell
Keywords: chronic lymphocytic leukemia; ibrutinib; arsenic trioxide; phosphatidylinositol 3-kinase
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Arsenic Trioxide; ibrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ibrutinib combined with As2O3 (Experimental): Ibrutinib combined with As2O3
  Interventions: Drug: Ibrutinib combined with As2O3
- Ibrutinib (Active Comparator): Ibrutinib only
  Interventions: Drug: ibrutinib

INTERVENTIONS:
Drug: Ibrutinib combined with As2O3 — arsenic trioxide combined with ibrutinib in CLL
  Other Names: Ibrutinib combined with arsenic trioxide
  Arms: Ibrutinib combined with As2O3
Drug: ibrutinib — ibrutinib
  Other Names: BTK inhibitor
  Arms: Ibrutinib

SUMMARY:
The purpose of this study is to determine whether the combination of As2O3 and ibrutinib is synergistic in chronic lymphocytic leukemia

DETAILED DESCRIPTION:
Chronic lymphocytic leukemia (CLL) is a common adult leukemia characterized by the extensive accumulation of monoclonal, relatively mature , positives of cluster of differentiation antigen 5 and cluster of differentiation antigen 23 B lymphocytes in lymphoid organs, bone marrow, and peripheral blood. CLL cells accumulate because of defective apoptosis, which extends survival. CLL is a heterogeneous disease. Chemoimmunotherapy is the standard front-line approach for patients younger than 65 years with CLL, with the combination of fludarabine, cyclophosphamide, and rituximab used most commonly. Some CLL patients do not respond well to routine chemoimmunotherapy. Despite recent advances in the treatment of CLL by use of modern chemoimmunotherapy, the disease remains incurable for most patients with the exception of those who have the option of an allogeneic transplantation. However, treatments with chemoimmunotherapy are associated with significant toxicities and sustained immunosuppression, and the rates of myelosuppression and infection are high. Such complications are more frequent and more severe in patients older than 65 years because of reduced marrow reserve, and presence of comorbidities. Because CLL is a disease of the elderly, identifying effective therapies with better toxicity profiles is thus a high priority, and targeted therapies may allow attainment of this goal.

Ibrutinib is an irreversible inhibitor of Bruton tyrosine kinase (BTK) that binds covalently to the cysteine residue (C481) in the kinase domain. This inhibition has been shown in vitro to induce modest CLL cell apoptosis and to abolish proliferation and B-cell receptor (BCR) signaling. Clinical trial results with this agent have been outstanding, including an estimated 26-month progression-free survival (PFS) of 75% for patients with relapsed and refractory disease. Although PFS with ibrutinib is excellent, the overall response rate for this group of relapsed patients is only 71%, lagging behind the clinical benefit seen in 88% of patients because of lymphocytosis induced by this agent and all agents targeting the BCR pathway.

Nevertheless, the long-term safety for ibrutinib has not been established. Caution must be exercised for the development of resistant clones due to the persistence of the disease, because most patients treated with ibrutinib often have prolonged partial remissions. Moreover, about 2-5% of CLL patients will develop Richter's syndrome or transformation during the disease course and treatment. The rate of serious adverse events in patients who continued treatment for 1 year or longer was 43% in the first year of treatment and 32% after the first year. Within the first year of treatment, 8% patients discontinued therapy, while 6% discontinued therapy after the first year. Besides, considering that genetic mutations cause resistance to ibrutinib in CLL patients and altered signaling pathways are common mechanisms of resistance to single agents. It's expected to combine other agent with ibrutinib to obtain higher response in those CLL patients who have not obtained perfect effect and to relieve the toxicity from treatment of ibrutinib.

However, arsenic trioxide (As2O3) has attracted worldwide interest in the field of oncology because of its substantial anticancer activity in patients with acute promyelocytic leukemia (APL). Interestingly, a number of studies have revealed that As2O3 can induce apoptosis, not only in APL, but also in a wide variety of hematologic malignancies, including CLL, either as monotherapy or combined therapy. Investigators previous study has also suggested that As2O3 could induce CLL cells apoptosis, and could be an efficient therapeutic agent for CLL.

ELIGIBILITY:
Inclusion Criteria:

* patients fulfilling clinical and immune-phenotypic criteria for CLL

Exclusion Criteria:

* none

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2016-12; Primary Completion 2017-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
overall response rate | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Xiao-Jun Huang, Doctor, Principal Investigator — Peking University People's Hospital

IPD SHARING:
Plan to Share IPD: Undecided